CLINICAL TRIAL: NCT03639896
Title: Endothelial Injury Mechanism of Cognitive Decline and Intervention Study in Elderly Patients Undergoing Major Surgery
Brief Title: Endothelial Injury Mechanism in Elderly Patients Undergoing Major Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Collaborators: Hangzhou Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7742
Record Dates: First submitted 2018-08-13; First posted 2018-08-21 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2019-09

CONDITIONS: Endothelial Dysfunction; Blood Brain Barrier Defect; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): 0.5μg/kg Dexmedetomidine as initial loading dose is given for 15 minutes before induction of anesthesia, followed by a maintenance infusion of 0.4μg/kg/h and stopped 30 minutes before the surgery over.
  Interventions: Drug: Dexmedetomidine
- Controlled (Placebo Comparator): 0.5μg/kg Saline as initial loading dose is given for 15 minutes before induction of anesthesia, followed by a maintenance infusion of 0.4μg/kg/h and stopped 30 minutes before the surgery over.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — 0.5μg/kg Dexmedetomidine as initial loading dose is given for 15 minutes before induction of anesthesia, followed by a maintenance infusion of 0.4μg/kg/h and stopped 30 minutes before the surgery over.
  Arms: Dexmedetomidine
Drug: Saline — 0.5μg/kg saline as initial loading dose is given for 15 minutes before induction of anesthesia, followed by a maintenance infusion of 0.4μg/kg/h and stopped 30 minutes before the surgery over.
  Arms: Controlled

SUMMARY:
The incidence of postoperative cognitive injury is high in elderly patients, especially after major surgery. The relevant pathophysiological mechanisms are still unclear, and the possible mechanisms that have been proposed so far include inflammation, neurotransmitter imbalance and metabolic disorders. In recent years, clinical studies of acute brain dysfunction after vascular endothelial injury have attracted attention.

Degradation of the endothelial glycocalyx layer and subsequent shedding of its constituents is seen as an early marker of endothelial injury, and may increase vascular permeability.Many preclinical and clinical studies have demonstrated an association between inflammatory cytokines such as TNF-α, IL-1β, IL-6, and IL-10 and glycocalyx degradation biomarkers.

The scholars found evidence of plasma endothelial injury after abdominal open surgery in the elderly. Dexmedetomidine could attenuate stress response such as TNF-α, IL-1β and IL-6. Based on the above evidence, we hypothesize that elderly patients experience inflammatory response secondary to surgical traumatic stress after major surgery, greatly increasing the degree of endothelial injury (heparan sulphate and syndecan-1), reducing brain perfusion while increasing Blood-brain barrier permeability (S100B level), promoting the release of cytokines Interleukin-2(IL-2), Interleukin-6(IL-6), tumor necrosis factor-alpha(TNF-α) ,and vascular endothelial growth factor (VEGF) while reducing brain-derived neurotrophic factor(BDNF) synthesis, then leading to postoperative acute spasm. We would test the hypothesis that can reverse these effects and improve cognitive deficits.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. Patients undergoing selective major gastrointestinal surgery with laparoscope and general anesthesia;
3. Age 65-90 yrs;
4. Anesthesia Society of American (ASA) Scale II~IV;
5. Anticipated surgery time 2-6 hrs;

Exclusion Criteria:

1. Dementia patients（Mini-mental state examination< 20）
2. Factors existed that affect cognition assessment such as language,visual,and auditory dysfunction；
3. Unstable metal status and mental disease；
4. A hematocrit value less than 28%in perioperative period;
5. Patients with abnormal preoperative inflammatory indicators（Higher white blood cell and C-reactive protein);
6. Patients undergoing cardiac and neural surgery;
7. Parkinson's Disease；
8. Sure or suspected abuse of analgesic and sedation drug.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 464 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
The change of incidence of postoperative delirium | The 1st, 2nd and 7th day after the surgery.
  Through CAM-ICU to assess the incidence of the postoperative delirium.
The change of incidence of postoperative cognition dysfunction | 1 day Before surgery,the 3rd,7th day after the surgery.
  The neuropsychological tests performed at the day before the surgery, the 3rd and 7th day after the surgery respectively.Calculate the difference(ΔX) between the score obtained before surgery and 3 or 7 days after the surgery (there are both positive and negative, we use the absolute value), with this difference( ΔX) divided by the standard deviation（SD）of the difference of the normal population, that is ΔX / SD and it is the Z score.If a patient has two or more than two of the absolute value of Z scores ≥1.96, the postoperative cognition dysfunction(POCD) is exist.

SECONDARY OUTCOMES:
endothelial injury levels | 1 day Before surgery,the 1st, 2nd, 3rd,7th day after the surgery.
  Plasma of patients was collected to test heparan sulphate and syndecan-1.
Blood-brain barrier permeability | 1 day Before surgery,the 1st, 2nd, 3rd,7th day after the surgery.
  Plasma of patients was collected to test S100B level
The serum concentrations of BDNF | 1 day Before surgery,the 1st, 2nd, 3rd,7th day after the surgery.
  Serum level of brain-derived neurotrophic factor (BDNF) was measured.
Inflammatory factor | 1 day Before surgery,the 1st, 2nd, 3rd,7th day after the surgery.
  Plasma of patients was collected to test cytokines IL-2, IL-6, TNF-α and VEGF level.

CONTACTS AND LOCATIONS:
Overall Officials: Xinqi Cheng, PhD, Principal Investigator — The First Affiliated Hospital of Anhui Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Hangzhou cancer hospital, Hangzhou, Zhejiang